CLINICAL TRIAL: NCT04118465
Title: Prospective Randomized Controlled Trial Comparing ECV Success Rates With and Without Full Urinary Bladder
Acronym: ECVBLADDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ezra Yosi, Director of Medical Unit, OB/GYN, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECVBLAD-HMO-CTIL
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Breech Presentation; Before Labor
Keywords: breech; ECV; version
MeSH Terms: conditions — Breech Presentation | interventions — Version, Fetal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECV with Full urinary bladder (Active Comparator): ECV with Full urinary bladder
  Interventions: Procedure: external cephalic version
- ECV with empty urinary bladder (Active Comparator): ECV with empty urinary bladder
  Interventions: Procedure: external cephalic version

INTERVENTIONS:
Procedure: external cephalic version — external cephalic version

SUMMARY:
A comparison of external cephalic (ECV) success rates when ECV performed with full urinary bladder or not. The study is prospective and randomised. Both nulliparous and multiparous women will be enrolled in the study, however each group will be randomized separately either to full urinary bladder or not. Written informed consent will be obtained prior to inclusion in the study.

DETAILED DESCRIPTION:
A comparison of external cephalic (ECV) success rates when ECV performed with full urinary bladder or not. The study is prospective and randomised. Both nulliparous and multiparous women will be enrolled in the study, however each group will be randomized separately either to full urinary bladder or not. Written informed consent will be obtained prior to inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* non-cephalic presentation,
* singleton pregnancy,
* term gestation,
* No previous attempt at ECV in this pregnancy,
* signed informed consent.

Exclusion Criteria:

• Any contraindication for vaginal delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 70 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ECV success rate | immediate
  ECV success rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion and publishing
Access Criteria: IPD will be supplied to interested research colleagues.

REFERENCES:
- [Derived] Kabiri D, Haj Yahya R, Yahalomi S, Ezra Y. Impact of full vs empty urinary bladder on external cephalic version success: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Jul;5(7):100991. doi: 10.1016/j.ajogmf.2023.100991. Epub 2023 Apr 30. PMID 38236701